CLINICAL TRIAL: NCT04323748
Title: The Use of Dose Dense Rituximab for High Risk Patients With Newly Diagnosed Acute Immune Thrombocytopenic Purpura
Brief Title: Dose Dense Rituximab for High Risk Newly Diagnosed Acute Immune Thrombocytopenic Purpura
Acronym: NYMC207
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14124
Record Dates: First submitted 2020-02-14; First posted 2020-03-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- rituximab (Experimental): All patients enrolled will receive the dose dense administration of rituximab. Five total doses will be administered on Days: 0, 2, 7 (± 2 days), 14 (± 2 days), and 21 (± 2 days); Dose: 375 mg/m2
  Interventions: Drug: rituxan

INTERVENTIONS:
Drug: rituxan — The dose dense administration of rituximab will consist of 5 doses total
  Days: 0, 2, 7 (± 2 days), 14 (± 2 days), and 21 (± 2 days); Dose: 375 mg/m2
  Other Names: rituximab

SUMMARY:
The purpose of this study is to determine if a dose dense administration of Rituximab in newly diagnosed acute immune thrombocytopenic purpura (ITP) and determine relapse rate following this treatment.

Correlative studies will be performed as outlined in the appendices.

Quality of Life will be measured using the KIT as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age: Subjects must be ≥ 1 year and ≤ 21 years of age.
* Diagnosis: Patients must have newly diagnosed ITP and a platelet count of ≤ 20 x 109 per Liter. Bone marrow aspirate and biopsy should be performed to rule out malignancy in the bone marrow.
* High-risk features : In addition, patients must have one of more of the following high-risk criteria:

  * Age ≥ 10 years
  * Grade II-IV bleeding at diagnosis
  * ANA positivity
  * No history of preceding infection within 2 weeks prior to ITP diagnosis
* Performance Status: Patients must have a performance status ≥ 50%. Use Karnofsky for patients > 16 years of age and Lansky for patients less than or equal to 16 years of age. See Appendix I for performance score.
* Prior Therapy

  * Patients may not have received any treatment for ITP prior to start of therapy.
  * Patients may not receive systemic steroids ≥ 0.5 mg/kg prednisone (or equivalent) within 2 weeks prior to diagnosis.
* Concomitant Medications Restrictions:

  * Steroids are only warranted as premedication prior to rituximab.
  * Patients who receive thrombopoetic agonists, eltrombopag or romiplostim will be taken off protocol.
* Organ Function Requirements

  * Adequate Renal Function Defined As: estimated CrCl > 60 mL/min or >30% of GFR for age based on the Schwartz formula
  * Adequate Liver Function Defined As: AST and/or ALT less than 5 times the upper limit of normal, and/or direct bilirubin less than the 2 times of the upper limit of normal

Exclusion Criteria

* Patients with a history of Grade III-IV allergic reaction to rituximab
* Patients with bone marrow neoplastic infiltration
* Patients with a history of hepatitis B infection
* Pregnancy and Breast Feeding

  * Female patients who are pregnant are ineligible (insert the reason: "due to risks of fetal and teratogenic adverse events as seen in animal/human studies" or "since there is yet no available information regarding human fetal or teratogenic toxicities").
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants.
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine the safety events: Number of participants with treatment-related Grade III or higher adverse events as assessed by CTCAE v5.0. | 1 year
  To determine the occurrence of any Grade ≥ 3 non hematologic toxicity (per CTCAE v.5) which is possibly, probably, or definitely related to rituximab.
To determine the Response Rate | 1 year
  To quantify remission rates for high-risk patients with acute ITP treated with a dose dense administration of rituximab.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Milner, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No